CLINICAL TRIAL: NCT05536414
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-arm Trial to Assess the Efficacy, Safety, and Tolerability of Centanafadine Extended-release Capsules as Monotherapy or as Adjunct to SSRI in Adult Subjects With Major Depressive Disorder
Brief Title: Trial of Centanafadine Efficacy and Safety as Monotherapy or as Adjunct to SSRI in Adults With Major Depressive Disorder
Acronym: JUNIPER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 405-201-00062
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder
Keywords: MDD; Centanafadine; SSRI; Depressive Disorder; Depression; Depressive Disorder, Major; Mood Disorders; Mental Disorders; Behavioral Symptoms
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder; Depression; Mood Disorders; Mental Disorders; Behavioral Symptoms | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Centanafadine + Placebo (Experimental)
  Interventions: Drug: Centanafadine; Drug: Placebo
- Centanafadine + Escitalopram (Experimental)
  Interventions: Drug: Centanafadine; Drug: Escitalopram
- Escitalopram + Placebo (Active Comparator)
  Interventions: Drug: Escitalopram; Drug: Placebo
- Placebo + Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Centanafadine — capsule
  Arms: Centanafadine + Escitalopram; Centanafadine + Placebo
Drug: Escitalopram — capsule
  Arms: Centanafadine + Escitalopram; Escitalopram + Placebo
Drug: Placebo — capsule
  Arms: Centanafadine + Placebo; Escitalopram + Placebo; Placebo + Placebo

SUMMARY:
This is a phase 2, multicenter, randomized, double-blind, placebo-controlled, parallel-arm trial to assess the efficacy, safety, and tolerability of centanafadine once-daily (QD) extended-release (XR) capsules for the treatment of adult subjects diagnosed with Major Depressive Disorder (MDD).

The trial will evaluate the efficacy and safety of centanafadine QD XR capsules as monotherapy or as adjunct to the selective serotonin reuptake inhibitor (SSRI), escitalopram.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and Female subjects between 18-65 years of age, with a primary diagnosis of major depressive disorder and in a current major depressive episode.
* History of an inadequate response to at least 1 and no more than 3 antidepressant treatments in the current major depressive episode.

Key Exclusion Criteria:

* Subjects who report an inadequate response to more than 3 antidepressant treatments in the current episode.
* Subjects with a lifetime history of schizophrenia spectrum or other psychotic disorder, bipolar or related disorder, neurocognitive disorder, or personality disorder.
* Subjects with a current diagnosis of post-traumatic stress disorder, obsessive compulsive disorder, panic disorder, or eating disorder (including anorexia nervosa or bulimia).
* Sexually active subjects, who could become pregnant, not agreeing to practice 2 sponsor approved methods of birth control or remain abstinent during the trial and for 30 days (females) or 90 days (males) after last dose of study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Week 6 in Montgomery-Asberg Depression Rating Scale (MADRS) Total score. | Baseline, Week 6

CONTACTS AND LOCATIONS:
Locations (62):
- United States (62):
  - Yuma CNS Research, Yuma, Arizona
  - SanRo Clinical Research Group LLC, Bryant, Arkansas
  - Behavioral Research Specialists-California-Irvine, Glendale, California
  - Sunwise Clinical Research, LLC - Lafayette - IVY - PPDS, Lafayette, California
  - OM Research LLC - Lancaster - ClinEdge - PPDS, Lancaster, California
  - Synergy Research Centers - SRC - ERG - PPDS, Lemon Grove, California
  - ATP Clinical Research, Orange, California
  - NRC Research Institute - Orange - PPDS, Orange, California
  - Prospective Research Innovations, Rancho Cucamonga, California
  - Anderson Clinical Research - ClinEdge - PPDS, Redlands, California
  - Lumos Clinical Research, San Jose, California
  - Syrentis Clinical Research, Santa Ana, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Viking Clinical Research Ltd, Temecula, California
  - CNS Clinical Research Group, Coral Springs, Florida
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Clinical Neuroscience Solutions Inc, Jacksonville, Florida
  - South Florida Research Phase I - IV, Miami Springs, Florida
  - Behavioral Clinical Research, Inc, North Miami, Florida
  - Clinical Neuroscience Solutions Inc, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Atlanta Center for Medical Research - CenExel ACMR - PPDS, Atlanta, Georgia
  - iResearch Atlanta - CenExel - PPDS, Decatur, Georgia
  - Psych Atlanta, Marietta, Georgia
  - Accelerated Clinical Trials,LLC, Peachtree Corners, Georgia
  - Northwest Clinical Trials, Boise, Idaho
  - Flourish Research - Andersonville - PPDS, Chicago, Illinois
  - Revive Research Institute, Elgin, Illinois
  - American Medical Research Inc, Oak Brook, Illinois
  - Louisiana Clinical Research, LLC, Shreveport, Louisiana
  - MTP Psychiatry, LLC, Baltimore, Maryland
  - Precise Research Centers - ClinEdge - PPDS, Flowood, Mississippi
  - Psychiatric Care and Research Center, O'Fallon, Missouri
  - Bio Behavioral Health, Toms River, New Jersey
  - Integrative Clinical Trials - Hunt - PPDS, Brooklyn, New York
  - SPRI Clinical Trials, LLC - ERG - PPDS, Brooklyn, New York
  - Fieve Clinical Research, New York, New York
  - Manhattan Behavioral Medicine, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Patient Priority Clinical Sites LLC, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Charak Clinical Research Center, Garfield Heights, Ohio
  - Neuro-Behavioral Clinical Research Inc - ClinEdge - PPDS, North Canton, Ohio
  - Cutting Edge Research, Oklahoma City, Oklahoma
  - Summit Research Network, Inc. - Portland - Headlands - PPDS, Portland, Oregon
  - Suburban Research Associates - ATLAS - West Chester - PPDS, West Chester, Pennsylvania
  - LLM Research - South Carolina, Myrtle Beach, South Carolina
  - Clinical Neuroscience Solutions Inc, Memphis, Tennessee
  - FutureSearch Trials of Dallas, LLC - IVY - PPDS, Dallas, Texas
  - InSite Clinical Research, LLC, DeSoto, Texas
  - Houston Mind & Brain, Houston, Texas
  - Innovative Medical Research of Texas, Houston, Texas
  - Red Oak Psychiatry Associates P A, Houston, Texas
  - University Hills Clinical Research, Irving, Texas
  - AIM Trials, Plano, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Alpine Research Organization, Inc, Clinton, Utah
  - Cedar Clinical Research - IVY - PPDS, Draper, Utah
  - The Memory Clinic, Bennington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Core Clinical Research, Everett, Washington

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com